CLINICAL TRIAL: NCT05827341
Title: A Real-World Study of COVID-19 Infection in Patients With Malignant Lymphomas Participating in Clinical Trials
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhiming, Prof., Sun Yat-sen University
Other Study IDs: B2023-075-01
Record Dates: First submitted 2023-04-22; First posted 2023-04-25 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Malignant Lymphoma; Clinical Trial; COVID-19
MeSH Terms: conditions — Lymphoma; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention needed

SUMMARY:
This study focuses on the population of malignant lymphoma patients who are also in clinical research. Through a real world cross-sectional survey of infection and death risk during the COVID-19 pandemic in Guangzhou from December 2022 to January 2023, this study aims to clarify the risk, level and mortality of lymphoma patients infected with COVID-19 during their clinical research, and provide necessary research data for Chinese lymphoma patients during the COVID-19 pandemic,

ELIGIBILITY:
Inclusion Criteria:

(1) the diagnosis of lymphoma was confirmed by pathology according to World Health Organization (WHO)-criteria; (2) diagnosed with COVID-19 based on a positive polymerase chain reaction (PCR) test result for SARS-CoV-2 from oropharyngeal swabs, or on a positive detection of covid-19 antigen from nasopharyngeal swabs and typical clinical history; (3) participated in registered clinical trials and received anti-lymphoma treatment within four weeks before COVID-19 infection; (4) complete data on clinico-pathological characteristics, treatment approaches and follow-up were available.

Exclusion Criteria:

* Patients who could not provide detailed information about COVID-19 infection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study focuses on the population of malignant lymphoma patients who are also in clinical research. Through a real world cross-sectional survey of infection and death risk during the COVID-19 pandemic in Sun Yat-Sen University Cancer Center from December 2022 to January 2023, this study aims to clarify the risk, level and mortality of lymphoma patients infected with COVID-19 during their clinical research, and provide necessary research data for Chinese lymphoma patients during the COVID-19 pandemic. We also aimed to identify risk factors of moderate/severe COVID-19 infection and hospital admission.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
The severity of COVID-19 | 2 months
  The severity of COVID-19 infection in maligant lymphoma patients evaluated by investigators
Hospital admission rate of COVID-19 infection | 2 months
  The percentage of malignant lymphoma patients who were admitted into hospital

CONTACTS AND LOCATIONS:
Overall Officials: Zhiming Li, Principal Investigator — Sun Yat-sen University
Locations (1):
- Department of Medical Oncology, Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No